CLINICAL TRIAL: NCT03092193
Title: Clinical Pharmacokinetics of Cytochrome P450: Influence on the Pharmacokinetics of Naproxen (CYP2C8 and CYP2C9) and Associated Naproxen-esomeprazole (CYP2C19)
Brief Title: Pharmacogenetic and Pharmacokinetics of Naproxen and Associated Naproxen-esomeprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriana Maria Calvo, Principal Investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 49806115.0.0000.5417
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Poor Metabolizer Due to Cytochrome P450 CYP2C9 Variant; Poor Metabolizer Due to Cytochrome p450 CYP2C19 Variant
Keywords: Naproxen; Association of naproxen-esomeprazole; High pressure liquid chromatography; Cytochrome P450
MeSH Terms: interventions — Naproxen; Cytochrome P-450 CYP2C9; Cytochrome P-450 CYP2C19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naproxen (Experimental): 20 patients will receive naproxen (one tablet 500 mg) to collected saliva samples for pharmacokinetic and pharmacogenetic studies
  Interventions: Drug: Naproxen
- Naproxen-esomeprazole (Experimental): 20 patients will receive after one month of first collection (with naproxen 500 mg), naproxen-esomeprazole (one tablet 500mg+20mg) to collected saliva samples for pharmacokinetic and pharmacogenetic studies
  Interventions: Drug: Naproxen-esomeprazole

INTERVENTIONS:
Drug: Naproxen — 20 phenotyped for CYP2C9 and CYP2C19 (by PCR) and for the pharmacokinetics of naproxen, saliva samples will be collected of these patients at different times after ingestion of a tablet of naproxen (500mg) (before, 0,25; 0,5; 0,75; 1; 1,5; 2; 3; 4; 5; 6; 8; 11; 24; 48; 72 e 96 hours after ingestion).
  Other Names: CYP2C9
  Arms: Naproxen
Drug: Naproxen-esomeprazole — 20 phenotyped for CYP2C9 and CYP2C19 (by PCR) and for the pharmacokinetics of naproxen-esomeprazole, saliva samples will be collected of these patients at different times after ingestion of a tablet of naproxen-esomeprazole (500mg+20mg) (after one month of the first collection) (before, 0,25; 0,5; 0,75; 1; 1,5; 2; 3; 4; 5; 6; 8; 11; 24; 48; 72 e 96 hours after ingestion).
  Other Names: CYP2C9; CYP2C19
  Arms: Naproxen-esomeprazole

SUMMARY:
The family of cytochrome P450 (CYP) is the most important drug metabolizing enzymes which contributes to the metabolism of a large proportion of drugs in humans. Some CYP450 enzymes reduce or alter the pharmacodynamic activity of many drugs and are involved in oxidative metabolism and elimination of many drugs commonly used by the population. Polymorphisms in CYP2C8 and CYP2C9 are common in different populations around the world and genetic variations in these alleles can cause decreased enzyme activity to nonsteroidal anti-inflammatory drugs (NSAIDs) such as celecoxib, diclofenac, ibuprofen, indomethacin, lornoxicam, meloxicam, valdecoxib, piroxicam, tenoxicam and naproxen. This compromise the bioavailability of the drug can alter the pharmacokinetics of these drugs and patients with mutations in these genes can exhibit increased plasma concentrations of values and areas under the curve (AUC), in addition to decreased clearance of drugs. Associations between NSAIDs and gastric protectors or proton pump inhibitors (PPIs) have become common nowadays, especially in patients who make chronic use of these drugs. Naproxen associated to esomeprazole, a proton pump inhibitor (PPI), was launched in the market recently and its application in acute pain is not yet elucidated. Esomeprazole suffers strong influence of CYP2C19 (hepatic drug-metabolizing enzyme that degrades PPIs). In patients with high enzyme activity of the CYP2C19, the drug can suffer high enzymatic degradation, and its diminished effect. Moreover, in patients with low enzyme CYP2C19 activity, the effect of acid inhibition by PPIs can be very strong.

DETAILED DESCRIPTION:
The genotype presented by the patient in relation to CYP2C8, 2C9 and 2C19 could influence the absorption and metabolism of these NSAIDs with or without the gastric protectors, and may differ from anti-inflammatory action and side effects. In this proposal, 20 volunteers will be genotyped and phenotyped for these haplotypes of cytochrome P450. For analysis of the proposed genes, saliva will be collected as a source of genomic DNA. For molecular analysis will be performed polymerase chain reaction (PCR) assays are used produced and validated by Applied Biosystems®. For pharmacokinetics will be collected saliva samples at various times after ingestion of a tablet of naproxen (500 mg) or naproxen associated to esomeprazole (500 + 20 mg), using mass spectrometry for analysis of drug concentrations in the samples. The results will be described with a 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Absence of infection and inflammation
* Absence of systemic diseases

Exclusion Criteria:

* patients with systemic diseases;
* patients with inflammation or infection;
* patients with a history of gastrointestinal bleeding or ulcerations;
* patients with cardiovascular, renal or hepatic diseases;
* patients who use antidepressant drugs, diuretics or anticoagulants;
* patients with a history of allergy to naproxen (500 mg);
* patients with a history of allergy to naproxen and ezomeprazole (500 mg and 20 mg);
* patients with a history of allergy to any other NSAID;
* pregnant and lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Saliva concentration of naproxen | one week after the ingestion
  20 phenotyped for CYP2C9 (by PCR) and for the pharmacokinetics of naproxen and naproxen-ezomeprazole saliva samples will be collected of these patients at different times after ingestion of a tablet of naproxen (500mg) (before, 0,25; 0,5; 0,75; 1; 1,5; 2; 3; 4; 5; 6; 8; 11; 24; 48; 72 e 96 hours after ingestion).
Saliva concentration of naproxen-esomeprazole | one week after ingestion
  20 phenotyped for CYP2C9 and CYP2C19 (by PCR) and for the pharmacokinetics of naproxen and naproxen-ezomeprazole saliva samples will be collected of these patients at different times after ingestion of a tablet of naproxen-esomeprazole (500mg+20mg) (before, 0,25; 0,5; 0,75; 1; 1,5; 2; 3; 4; 5; 6; 8; 11; 24; 48; 72 e 96 hours after ingestion).

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Calvo, PhD, Study Chair — Bauru School of Dentistry/USP
Locations (1):
- Bauru School of Dentistry/USP, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No